CLINICAL TRIAL: NCT04252469
Title: Efficacy of Pre-intubation Chlorhexidine Oral Care on Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201806086RINB
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Intratracheal Intubation; Surgery; Anesthesia
Keywords: oral care; Anesthesia; surgery; Intratracheal Intubation
MeSH Terms: interventions — Dental Care Team

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): receiving oral care with 20mL of 0.12% CHX by medicine cup, gargling 30 seconds.
  Interventions: Other: Oral care
- Control (No Intervention): Standardized care

INTERVENTIONS:
Other: Oral care — oral care using 20mL of 0.12% CHX and gargling with 30 seconds.
  Arms: intervention

SUMMARY:
This single-centre, single-blind, randomised controlled study with parallel-group design was conducted in Yun Ling, Taiwan between May 2019 and August 2019. Participants were randomly allocated to an intervention (mouth care using 0.12% CHX before intubation) or control (standard care) group on a 1:1 basis. This study was approved by the institutional review board of National Taiwan University Hospital, Taiwan (IRB No.201806086RINB). Each participant completed written informed consent after explanation of this study and advised that they could withdraw anytime.

DETAILED DESCRIPTION:
Participants were recruited at the operation room of a teaching hospital. Participants were included if they met the following criteria: 18-80 years of age, American Society of Anesthesiologists, ASA) class 1-3, scheduled for surgery under endotracheal tube intubation general anesthesia. Patients were excluded if they were diagnosed with upper or lower respiratory tract disease, including COPD, cold, had oral ulcer, scheduled to have a respiratory-related surgical procedure, had endotracheal tube intubated.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, American Society of Anesthesiologists, ASA) class 1-3, scheduled for surgery under endotracheal tube intubation general anesthesia.

Exclusion Criteria:

* Patients were excluded if they were diagnosed with upper or lower respiratory tract disease, including COPD, cold, had oral ulcer, scheduled to have a respiratory-related surgical procedure, had endotracheal tube intubated, >1 during anesthesia processes,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Bacterial Colonization (Gram stain) | at baseline (30 minutes before surgery started)
  Bacterial Colonization
Bacterial Colonization (Gram stain) | at removal of endotracheal tube (3 minutes after surgery ended and removal of endotracheal tube )
  Bacterial Colonization
Bacterial Colonization (Gram stain) | after removal of endotracheal tube at recovery room (15 minutes after surgery ended)
  Bacterial Colonization

SECONDARY OUTCOMES:
Breathing odor assessment using questionnaire | at baseline (30 minutes before surgery started)
  Breathing odor assessment
Breathing odor assessment using questionnaire | at insertion of endotracheal tube
  Breathing odor assessment
Breathing odor assessment using questionnaire | after removal of endotracheal tube and at recovery room (15 minutes after surgery ended)
  Breathing odor assessment
Breathing odor assessment using halitosis detector | at baseline (30 minutes before surgery started)
  Breathing odor assessment
Breathing odor assessment using halitosis detector | after removal of endotracheal tube and at recovery room (15 minutes after surgery ended)
  Breathing odor assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wyee Lee, MSN, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricard JD, Lisboa T. Caution for chlorhexidine gluconate use for oral care: insufficient data. Intensive Care Med. 2018 Jul;44(7):1162-1164. doi: 10.1007/s00134-018-5217-6. Epub 2018 May 15. No abstract available. PMID 29766214
- [Result] Deschepper M, Waegeman W, Eeckloo K, Vogelaers D, Blot S. Effects of chlorhexidine gluconate oral care on hospital mortality: a hospital-wide, observational cohort study. Intensive Care Med. 2018 Jul;44(7):1017-1026. doi: 10.1007/s00134-018-5171-3. Epub 2018 May 9. PMID 29744564
- [Result] La Combe B, Maherault AC, Messika J, Billard-Pomares T, Branger C, Landraud L, Dreyfuss D, Dib F, Massias L, Ricard JD. Oropharyngeal Bacterial Colonization after Chlorhexidine Mouthwash in Mechanically Ventilated Critically Ill Patients. Anesthesiology. 2018 Dec;129(6):1140-1148. doi: 10.1097/ALN.0000000000002451. PMID 30247201